CLINICAL TRIAL: NCT06952348
Title: HYPERtension Reduction Through WALKing Stairs Versus Brisk Walking in Individuals With Increased Cardiometabolic Risk - The HYPERWALK Randomized Controlled Trial
Brief Title: HYPERtension Reduction Through WALKing Stairs Versus Brisk Walking
Acronym: HYPERWALK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Södersjukhuset (Stockholm South General Hospital) (Unknown); Ersta Cardiology Outpatient Clinic (Unknown); Liljeholmens vårdcentral (Unknown); Boo vårdcentral (Unknown); Karolinska University Hospital (Other); Sodertalje Hospital (Other)
Responsible Party: Principal Investigator, Pontus Andell, Associate Professor, Consultant in Cardiology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-05912-01
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Disease; Cardiovascular Diseases; Hypertension; Obesity and Overweight
Keywords: Cardiovascular prevention; Physical activity; Smart medicine; Obesity; Overweight; Hypertension
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases; Hypertension; Obesity; Overweight; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, participant blinding is not feasible. To ensure validity, group allocation will be disclosed only after baseline data collection and by personnel not involved in outcome assessments. To preserve assessor blinding at follow-up, participants will be instructed not to reveal their group assignment. Additionally, study staff will document whether blinding was maintained after each follow-up assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stair and brisk walking combined (Experimental): Participants will double their baseline physical activity levels by combining stair walking and brisk walking. The stair walking goal is ≥250 steps per day (equivalent to ~37.5-45 meters elevation or 15 floor levels), totaling ~37.5 minutes per week. In addition, they will complete ≥75 minutes of brisk walking per week.
  Interventions: Behavioral: Stair and brisk walking combined
- Brisk walking (Experimental): Participants will double their baseline physical activity levels by engaging in brisk walking only, with a minimum target of >150 minutes per week.
  Interventions: Behavioral: Brisk walking
- Standard care (Active Comparator): Participants will receive general lifestyle advice aligned with current physical activity guidelines but will not be provided with specific exercise instructions, personalized activity targets, or feedback. They will wear the same activity monitor as the intervention groups, but without access to feedback or goal-setting features.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Stair and brisk walking combined — See arms.
  Arms: Stair and brisk walking combined
Behavioral: Brisk walking — See arms.
  Arms: Brisk walking
Behavioral: Standard care — See arms.
  Arms: Standard care

SUMMARY:
This clinical trial investigates whether incorporating stair walking into daily routines improves physical health in adults at risk of lifestyle-related conditions such as hypertension, type 2 diabetes, and cardiovascular disease. Participants will be randomized into three groups: (1) stair walking combined with brisk walking, (2) brisk walking alone, and (3) a control group receiving standard lifestyle advice without specific exercise instructions, stratified by age (<65 y/o, v >=65) and site.

The primary objective is to assess whether the combination of stair and brisk walking leads to greater reductions in systolic blood pressure compared to brisk walking alone or standard care. Secondary outcomes include changes in cardiometabolic risk factors.

Participants in the stair walking group will be instructed to climb ≥250 steps per day (~5.5 minutes/day or ~37.5 minutes/week), or complete an equivalent elevation via inclined slopes, along with ≥75 minutes of brisk walking per week. Those in the brisk walking group will walk ≥150 minutes per week. The control group will receive general lifestyle advice but no tailored physical activity goals or feedback.

Participants in both active groups will aim to double their baseline activity levels. Physical activity will be continuously monitored using wearable devices. The active groups will receive personalized feedback and motivational support throughout the 6-month intervention period.

If effective, this study may offer a simple, scalable, and low-cost intervention model for use in clinical and public health settings, emphasizing personalized goals, remote monitoring, and behavioral support.

ELIGIBILITY:
Inclusion Criteria

Men and women aged 35 years or older with increased cardiometabolic risk, defined by all of the following:

1. Clinically confirmed hypertension, with or without antihypertensive treatment, as documented in the Electronic Health Record (EHR).
2. Overweight or obesity, defined as BMI between 27 and 40.
3. Physically inactive lifestyle, defined as either:

   * Light intensity or inactive category on the Stanford Brief Activity Survey (SBAS), or
   * Light intensity or inactive category in the physical activity section of the Swedish National Board of Health and Welfare Lifestyle Questionnaire.

Exclusion Criteria

Medical contraindications to physical activity (based on FYSS 2021, p. 182):

* Severe, symptomatic aortic stenosis
* Acute pulmonary embolism, myocarditis, pericarditis, or systemic infection (e.g., fever, muscle pain, lymphadenopathy)
* Suspected or known aortic dissection
* Severe hypertension (Grade 3: SBP >180 mmHg or DBP >110 mmHg), regardless of symptoms
* Unstable coronary artery disease (including unstable angina, suboptimally treated stable angina, or recent myocardial infarction <8 weeks)
* Symptomatic, uncontrolled arrhythmia
* Symptomatic, uncontrolled heart failure

Other exclusion criteria:

* Implanted pacemaker or ICD
* Pregnancy
* Smartphone incompatibility with Fitrockr© app (iOS <16 or Android OS <10)
* Inability to understand Swedish or English
* Any condition that may interfere with protocol compliance (e.g., severe mental illness or cognitive impairment)
* Inability to walk stairs

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) at 6 months | 6 months
  Office systolic blood pressure (SBP) at 6-month follow-up, adjusted for baseline values. SBP is a validated and widely accepted surrogate marker for cardiovascular morbidity and mortality, as well as overall health risk.

SECONDARY OUTCOMES:
Diastolic Blood Pressure (DBP) | 6 months
  Office diastolic blood pressure (DBP) at 6-month follow-up, adjusted for baseline values. DBP is a clinically relevant indicator of cardiovascular risk and contributes to the assessment of overall blood pressure control.
HOMA-index | 6 months
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at 6-month follow-up, adjusted for baseline values. HOMA-IR is a validated surrogate marker of insulin resistance and metabolic risk, commonly used in cardiometabolic research.
HbA1c | 6 months
  Hemoglobin A1c (HbA1c) at 6-month follow-up, adjusted for baseline values. HbA1c reflects average blood glucose levels over the preceding 2-3 months and is a standard marker for assessing glycemic control and diabetes risk.
LDL cholesterol | 6 months
  Low-Density Lipoprotein (LDL) cholesterol at 6-month follow-up, adjusted for baseline values. LDL cholesterol is a key biomarker for cardiovascular risk and a primary target in lipid-lowering therapies.
Triglycerides | 6 months
  Triglycerides (TG) at 6-month follow-up, adjusted for baseline levels. Elevated TG are associated with increased cardiovascular risk and are a core component of the metabolic syndrome.

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Liljeholmen Primary Care Center, Stockholm
  - Södersjukhuset, Stockholm
  - Södertälje sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Blood pressure (systolic and diastolic), BMI, sex, age, HOMA-index, HbA1c, Triglycerides, LDL will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT06952348/Prot_SAP_002.pdf